CLINICAL TRIAL: NCT01841268
Title: Skin Lipid Profiles in Term and Preterm Infants
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 240869
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Preterm Infants
Keywords: premature, preterm, premie, skin
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Blood, epidermal skin cells, breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm Infants: Infants born prematurely will have their skin, sebum, microbiota, blood, and mother's breast milk analyzed for changes between 0, 2, and 4 weeks of life.
- Term Infants, Control: Term infants enrolled in the UC Davis Lactation Study (protocol # 216198) will serve as the control group for this study; they will have their skin, sebum, microbiota, and mother's breast milk analyzed for changes between 0, 2, and 4 weeks of life.

SUMMARY:
This study is designed to compare the skin lipid and protein composition between term and premature infants and determine how the skin composition changes over the first four weeks of life. The investigators hope to elucidate the unique characteristics of premature skin by measuring the lipid and protein content in skin, how it changes during the first month of life, and how it varies with formula feeding versus breast feeding. Additionally, the investigators will study the relationships among diet, skin composition and plasma lipids in premature infants over the first four weeks of life.

DETAILED DESCRIPTION:
Infants in the UCDMC Neonatal Intensive Care Unit with no congenital or acquired diseases of the skin or cardiovascular system will be enrolled after informed consent has been obtained from their parents. This is an observational study with no intervention. Procedures: At enrollment, 2 weeks and 4 weeks of age, skin lipids will be collected using three methods. First two small pieces of blotting paper (2 cm x 2 cm) will be placed on the infant's skin, one on the left side of the abdomen just above the umbilicus and one on the left inner thigh. The blotting paper will be left in place for 15 seconds and then removed. Second, two adhesive discs will be placed on the skin, one just below the umbilicus and one on the right inner thigh. The discs will be left in place for 30 seconds and then removed. Third, two areas of skin, one on the right side of the abdomen just above the umbilicus and the other on the inner right thigh, will be gently swabbed with sterile cotton swabs (one for each location). The intent is to remove a thin layer of oil/lipid from the skin upon removal of the paper or the adhesive disc or with swabbing without disrupting the skin surface (similar to taking a fingerprint). Blood specimens will be obtained three times, each time 1 ml : once at enrollment, at 2 weeks and the last one at 4 weeks of age, to generate a plasma lipoprotein profile and size distribution (HDL, LDL, VLDL, total cholesterol). For infants that are fed expressed human milk, we will also obtain a sample of mother's milk for analysis of lipid profile (about 2 ml).

ELIGIBILITY:
Inclusion Criteria:

* infants who are likely to be inpatients in the NICU for at least 4 weeks

Exclusion Criteria:

* congenital or acquired skin disease,
* cyanotic congenital heart disease,
* neonates that are not viable and
* those with lethal anomalies such as anencephaly, trisomy 13, trisomy 18, renal agenesis

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn infants in the NICU at UCDMC. 20 neonates will be enrolled, 5 in each of the following gestational age categories: 23-27 weeks, 28-32 weeks, 33-36 weeks, >36 weeks. Infants will be involved in the study from enrollment until 4 weeks of age or until discharge, whichever comes first.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Skin Proteome | Change between 0, 2, and 4 weeks
  Premie infant skin proteome changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life.
Skin Lipidome | Changes between 0, 2, and 4 weeks
  Premie infant skin lipidome changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Skin Microbiota | Changes between 1, 2, and 4 weeks
  Premie infant skin microbiota changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Skin Sebum | Changes between 0, 2, and 4 weeks
  Premie infant skin sebum changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Breast Milk Lipidome | Changes between 0, 2, and 4 weeks
  Mothers of premie infants will have their breast milk lipidome analyzed for changes between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Breast Milk Fatty Acids | Changes between 0, 2, and 4 weeks
  Mothers of premie infants will have their breast milk fatty acids analyzed for changes between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Plasma Lipoprotein Profile(HDL, LDL, VLDL, total cholesterol) | Changes between 0, 2, and 4 weeks
  Premie infant lipoprotein (HDL, LDL, VLDL, total cholesterol) profile changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Plasma Lipoprotein Size Distribution(HDL, LDL, VLDL, total cholesterol) | Changes between 0, 2, and 4 weeks
  Premie infant lipoprotein (HDL, LDL, VLDL, total cholesterol) size distribution changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life
Plasma Fatty Acid Analysis | Changes between 0, 2, and 4 weeks
  Premie infant plasma fatty acid analysis changes will be determined between 0 weeks (less than 5 days of life), 2 weeks, and 4 weeks of life

CONTACTS AND LOCATIONS:
Overall Officials: Mark Underwood, M.D., Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California, Davis, Davis, California
  - University of California Davis Medical Center NICU, Sacramento, California

REFERENCES:
- [Background] Nilsson GE. Measurement of water exchange through skin. Med Biol Eng Comput. 1977 May;15(3):209-18. doi: 10.1007/BF02441040. No abstract available. PMID 195148
- [Background] Agren J, Sjors G, Sedin G. Ambient humidity influences the rate of skin barrier maturation in extremely preterm infants. J Pediatr. 2006 May;148(5):613-7. doi: 10.1016/j.jpeds.2005.11.027. PMID 16737871
- [Background] Jiang YJ, Barish G, Lu B, Evans RM, Crumrine D, Schmuth M, Elias PM, Feingold KR. PPARdelta activation promotes stratum corneum formation and epidermal permeability barrier development during late gestation. J Invest Dermatol. 2010 Feb;130(2):511-9. doi: 10.1038/jid.2009.245. Epub 2009 Aug 13. PMID 19675577
- [Background] Feingold KR, Schmuth M, Elias PM. The regulation of permeability barrier homeostasis. J Invest Dermatol. 2007 Jul;127(7):1574-6. doi: 10.1038/sj.jid.5700774. PMID 17568800
- [Background] Weerheim A, Ponec M. Determination of stratum corneum lipid profile by tape stripping in combination with high-performance thin-layer chromatography. Arch Dermatol Res. 2001 Apr;293(4):191-9. doi: 10.1007/s004030100212. PMID 11380152
- [Background] Holleran WM, Takagi Y, Uchida Y. Epidermal sphingolipids: metabolism, function, and roles in skin disorders. FEBS Lett. 2006 Oct 9;580(23):5456-66. doi: 10.1016/j.febslet.2006.08.039. Epub 2006 Sep 1. PMID 16962101
- [Background] Bennett K, Callard R, Heywood W, Harper J, Jayakumar A, Clayman GL, Di WL, Mills K. New role for LEKTI in skin barrier formation: label-free quantitative proteomic identification of caspase 14 as a novel target for the protease inhibitor LEKTI. J Proteome Res. 2010 Aug 6;9(8):4289-94. doi: 10.1021/pr1003467. PMID 20533828
- [Background] Rice RH, Rocke DM, Tsai HS, Silva KA, Lee YJ, Sundberg JP. Distinguishing mouse strains by proteomic analysis of pelage hair. J Invest Dermatol. 2009 Sep;129(9):2120-5. doi: 10.1038/jid.2009.52. Epub 2009 Mar 19. PMID 19295613
- [Result] Scoble JA, Smilowitz JT, Argov-Argaman N, German JB, Underwood MA. Plasma Lipoprotein Particle Subclasses in Preterm Infants. Am J Perinatol. 2018 Mar;35(4):369-379. doi: 10.1055/s-0037-1607347. Epub 2017 Oct 26. PMID 29076117
- [Derived] Spevacek AR, Smilowitz JT, Chin EL, Underwood MA, German JB, Slupsky CM. Infant Maturity at Birth Reveals Minor Differences in the Maternal Milk Metabolome in the First Month of Lactation. J Nutr. 2015 Aug;145(8):1698-708. doi: 10.3945/jn.115.210252. Epub 2015 Jun 3. PMID 26041675